CLINICAL TRIAL: NCT07155096
Title: Accelerated DMN-Targeted cTBS to Modulate DMN Connectivity
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Heather Burrell Ward, Principle Investigator, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 232140
Record Dates: First submitted 2025-08-26; First posted 2025-09-04 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Schizophrenia
Keywords: schizophrenia; rTMS; TMS; fMRI; DMN
MeSH Terms: conditions — Schizophrenia | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Default Mode Network-Targeted cTBS (Experimental): All participants receive 5 sessions of active cTBS (600 pulses) to the DMN, with a 30-minute inter-session interval.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — Repetitive Transcranial Magnetic Stimulation (rTMS): Participants will each receive Default Mode Network-targeted continuous theta burst stimulation (cTBS) administered at 100% Active Motor Threshold

SUMMARY:
The central hypothesis is this: DMN connectivity can be modulated with inhibitory cTBS when delivered on an accelerated treatment schedule. This study seeks to provide evidence that accelerated, network-targeted inhibitory stimulation of the DMN leads to both altered network activity and a concomitant behavioral change in cognitive performance in individuals with schizophrenia and schizoaffective disorder. This study will also compare the effect of inhibitory cTBS in healthy individuals, as it may also lead to both altered network activity and a behavioral change in cognitive performance in individuals without schizophrenia or schizoaffective disorder.

If successful, this study will have identified a safe, effective, and broadly applicable treatment for cognitive impairment in schizophrenia that has potential for translation into many other psychiatric and neurodevelopmental disorders, such as autism.

DETAILED DESCRIPTION:
Schizophrenia and other psychotic disorders are disabling, lifelong illnesses that afflict over three million people in the US. Schizophrenia is characterized by positive symptoms (i.e., delusions, hallucinations), negative symptoms (i.e., anhedonia, amotivation), and cognitive impairment. Cognitive impairment is a devastating, central and enduring feature of schizophrenia that is a leading cause of disability. Nearly 94% of people with schizophrenia have at least one cognitive symptom. However, there are no current treatments for cognitive impairment in schizophrenia.

DMN hyperconnectivity has been observed across multiple psychiatric disorders, including schizophrenia. DMN disruption in schizophrenia is a well-replicated observation. DMN disorganization has been consistently observed in individuals with schizophrenia and their first-degree relatives and has been associated with cognitive impairment, positive symptoms, negative symptoms, and nicotine use. Therefore, DMN connectivity may be a potential biomarker and treatment target for cognitive impairment across multiple psychiatric disorders, including schizophrenia and autism.

Repetitive transcranial magnetic stimulation (rTMS) is a form of non-invasive brain stimulation that uses electromagnetic fields to change neuronal patterns of connectivity in brain networks. When international safety guidelines are followed, rTMS is a safe and well-tolerated intervention in individuals with and without psychiatric illness (Rossi et al. 2021). rTMS is also a versatile research tool whose stimulation parameters can be changed. Depending on the parameters, rTMS can be excitatory or inhibitory and can increase or decrease network connectivity. Specifically, intermittent theta burst stimulation (iTBS) is excitatory, while continuous theta burst stimulation (cTBS) is inhibitory. In this protocol, inhibitory cTBS is used to reduce DMN connectivity and improve cognitive performance. rTMS has been successfully used to modulate DMN connectivity in healthy individuals and in individuals with psychosis. rTMS is FDA-approved for the treatment of major depressive disorder, obsessive-compulsive disorder, and smoking cessation.

Previous studies by our group and others have demonstrated the ability of rTMS to change patterns of activity in cortical networks of the human brain. In addition, researchers have also previously demonstrated the ability to both increase and decrease connectivity within a specific network (e.g. DMN) by neuroanatomically targeted rTMS. In the present study, an accelerated inhibitory cTBS intervention will be delivered to the left parietal node of the DMN, a network key to attentional performance. The PI has conducted clinical trials testing both single and multiple sessions of cTBS to the parietal node of the DMN. cTBS applied to the parietal cortex has been well tolerated, and there have been no serious adverse events, including no worsening of psychosis or depression, and no seizures. In fact, 5 sessions of DMN-targeted cTBS (which will be used in this study) significantly reduced nicotine craving in schizophrenia. cTBS has also been investigated as a treatment for seizures.

In most clinical and research protocols, rTMS is traditionally applied in daily sessions for 4-6 weeks. However, accelerated protocols have recently consolidated treatment into multiple rTMS sessions per day, thereby reducing treatment duration and shortening time to achieve clinical response. Accelerated protocols also offer significant advantages for other clinical populations, such as neurodevelopmental disorders, where daily treatment over multiple weeks may not be feasible. Currently, an FDA-cleared accelerated rTMS for depression involves treatment with 10 excitatory rTMS sessions/day for 5 days (i.e., 50 rTMS sessions over 1 week). In the current protocol, this study will test 5 inhibitory cTBS sessions delivered in 1 day.

Our central hypothesis is this: DMN connectivity can be modulated with inhibitory cTBS when delivered on an accelerated treatment schedule. This study seeks to provide evidence that accelerated, network-targeted inhibitory stimulation of the DMN leads to both altered network activity and a concomitant behavioral change in cognitive performance in individuals with schizophrenia and schizoaffective disorder. This study will also compare the effect of inhibitory cTBS in healthy individuals, as it may also lead to both altered network activity and a behavioral change in cognitive performance in individuals without schizophrenia or schizoaffective disorder.

If successful, this study will have identified a safe, effective, and broadly applicable treatment for cognitive impairment in schizophrenia that has potential for translation into many other psychiatric and neurodevelopmental disorders, such as autism.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-65 years
* Diagnosis of either schizophrenia or schizoaffective disorder according to DSM-5 criteria and confirmed by SCID (First et al. 2015)
* Must be able to read, speak and understand English
* Must be judged by study staff to be capable of completing the study procedures
* Participants will be in stable outpatient psychiatric treatment and psychiatrically stable with no recent (within the past 30 days) psychiatric hospitalizations or changes in their psychiatric medication regimens.

Exclusion Criteria:

* • DSM-5 intellectual disability

  * Substance use disorder (other than nicotine) within the past three months
  * Current, active suicidal ideation with intent or plan, as assessed by a score of 5 or higher on the Brief Psychiatric Rating Scale question #4 Suicidality.
  * Positive urine drug screen for illicit substance use that can increase seizure risk (cocaine, benzodiazepines, amphetamine, methamphetamine)
  * Any history of a progressive or genetic neurologic disorder (e.g. Parkinson's disease, multiple sclerosis, tuberous sclerosis, Alzheimer's Disease) or acquired neurological disease (e.g. stroke, traumatic brain injury, tumor), including intracranial lesions
  * History of head trauma resulting in any loss of consciousness (>15 minutes) or neurological sequelae
  * Current history of poorly controlled headaches including chronic medication for migraine prevention
  * History of fainting spells of unknown or undetermined etiology that might constitute seizures
  * History of seizures, diagnosis of epilepsy, or immediate (1st degree relative) family history epilepsy with the exception of a single seizure of benign etiology (e.g. febrile seizures) in the judgment of a board-certified neurologist
  * Chronic (particularly) uncontrolled medical conditions that may cause a medical emergency in case of a provoked seizure (cardiac malformation, cardiac dysrhythmia, asthma, etc.)
  * Any metal in the brain or skull (excluding dental fillings) or elsewhere in the body unless cleared by the responsible covering MD (e.g. MRI compatible joint replacement)
  * Any devices such as pacemaker, medication pump, nerve stimulator, TENS unit, ventriculo-peritoneal shunt unless cleared by the responsible covering MD
  * All female participants of child-bearing age will be required to have a pregnancy test; any participant who is pregnant or planning to become pregnant will not be enrolled in the study
  * Medications will be reviewed by the responsible covering physician and a decision about inclusion will be made based on the participant's past medical history, drug dose, history of recent medication changes or duration of treatment, and use of CNS active drugs. The published TMS guidelines review of medications to be considered with rTMS will be taken into consideration given their described effects on cortical excitability measures.
  * Any changes in medications or hospitalizations within the past 30 days.
  * Participants who, in the investigator's opinion, might not be suitable for the study or would be unable to tolerate the study visit

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09-09 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Functional Connectivity Changes | From enrollment to the end of MRI, maximum 3 weeks.
  We will determine if an accelerated inhibitory cTBS protocol targeted to the DMN is associated with a decrease in functional connectivity before and after cTBS

SECONDARY OUTCOMES:
Cognitive Performance | From enrollment to the end of the study, maximum 3 weeks.
  As an exploratory analysis, we will also determine if change in DMN functional connectivity is associated with change in cognitive performance.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Ward, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt Psychiatric Hospital, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
This study is not NIH-funded, so public data sharing is not required. Reasonable requests for data sharing will be considered.